CLINICAL TRIAL: NCT02370667
Title: Clinical and Tissue Outcomes of a Biomechanical Exercise Program for Knee Osteoarthritis
Brief Title: A Biomechanical Exercise Program for Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BiomechanicalExerciseProgram
Record Dates: First submitted 2015-02-09; First posted 2015-02-25 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Exercise; Magnetic Resonance Imaging
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Biomechanical Exercise (BE) (Experimental): The participants in this arm will be asked to attend 3 group classes per week for 12 weeks at a local yoga studio taught by a certified yoga instructor. Four class times will be offered per week. These classes will include a warm-up, static poses shown to decrease knee joint loading, and a cool down including flexibility exercises. Measurements will be obtained at baseline (before intervention) and at follow-up (following intervention). Outcomes will include clinical mobility; muscle and fat volumes, and cartilage morphology using MRI; pain; isometric leg strength; cardiovascular fitness; and gait analysis.
  Interventions: Other: Biomechanical Exercise (BE)
- Traditional Exercise (TE) (Active Comparator): The participants in this arm will be prescribed an aerobic and strengthening exercise program often prescribed to those with knee OA. The program will include 15 minutes of walking per class, closed kinetic chain strengthening exercises on machines, and a cool down consisting of stretching. Participants will be asked to come to class 3 times per week for 12 weeks. Certified Kinesiologists as well as student volunteers will be available during all class times for program completion and progression.
  Interventions: Other: Traditional Exercise (TE)
- Meditation Control (M) (Other): The participants in this arm will be asked to attend 3 meditation classes per week for 12 weeks taught by a certified yoga instructor with a specialization in meditation. This will take place at an alternate yoga studio to avoid contamination. Since it is known that exercise is beneficial for pain management and strengthening in knee OA, participants randomized to the control group will be offered a free exercise pass following completion of the study.
  Interventions: Other: Meditation Control (M)

INTERVENTIONS:
Other: Biomechanical Exercise (BE) — A biomechanical exercise program shown to decrease joint loading will be administered 3 times a week for 12 weeks. Outcomes will include mobility performance; pain; muscle and fat volumes, and cartilage morphology using MRI; strength; cardiovascular fitness; and gait analysis.
  Arms: Biomechanical Exercise (BE)
Other: Traditional Exercise (TE) — A traditional exercise program for people with knee OA will be administered 3 times a week for 12 weeks. Outcomes will include mobility performance; pain; muscle and fat volumes, and cartilage morphology using MRI; strength; cardiovascular fitness; and gait analysis.
  Arms: Traditional Exercise (TE)
Other: Meditation Control (M) — A meditation program acting as a control will be administered 3 times a week for 12 weeks. Outcomes will include mobility performance; pain; muscle and fat volumes, and cartilage morphology using MRI; strength; cardiovascular fitness; and gait analysis.
  Arms: Meditation Control (M)

SUMMARY:
Prescribing exercise for people with painful knee osteoarthritis (OA) is essential for pain management, improved function, and chronic disease prevention. Exercise that decreases joint exposure to damaging loading while eliciting adequate muscular activation for strength improvements is ideal. The purpose of this 3-arm RCT is to compare mobility, strength, pain, and MRI outcomes between the low-loading biomechanical exercise program (BE), a traditional exercise program for knee OA (TE), and a control group completing meditation classes (M).

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a common joint disease affecting 1 in 10 Canadians. Osteoarthritis commonly presents in the knee joint and is associated with mobility limitations, pain, and an increased risk of other chronic health conditions such as heart disease. It is critical to implement exercise for people with knee OA as it can be an effective method for improving pain, mobility, and cardiovascular health. A biomechanical exercise program using static yoga postures has been established in the investigators lab based on minimizing damaging knee joint loads, while effectively exercising the musculature around the knee joint. The investigators pilot project (REB#13-510) showed that a 12-week yoga program using these biomechanical exercises improved pain and mobility while keeping the medial joint loading well below that experienced during normal level walking. The next step with this exercise program is to compare clinical and tissue outcomes with that of a regularly prescribed aerobic and strengthening program, as well as a control group completing meditation classes. The investigators aim to identify differences in clinical mobility performance outcomes, muscle and fat volumes using magnetic resonance imaging (MRI), and cartilage integrity using MRI between the three groups using a randomized controlled trial (RCT) design.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older
* Knee pain on most days of the week
* Less than 30 minutes of morning stiffness
* Bony enlargement
* Bony tenderness to palpation
* Signs of inflammation
* Able to safely climb 2 flights of stairs without aid

Exclusion Criteria:

* Any other forms of arthritis
* Osteoporosis
* History of patellofemoral symptoms
* Active non-arthritic knee disease
* Knee surgery
* Use of cane or walking aid
* Unstable heart condition
* Neurological conditions
* Skin allergy to medical tape
* Hip or ankle injuries in past 3 months
* Any injuries that would prohibit participation in yoga
* Ipsilateral hip or ankle conditions
* Currently receiving cancer treatment
* Currently pregnant

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica R Maly, PT, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuntz AB, Chopp-Hurley JN, Brenneman EC, Karampatos S, Wiebenga EG, Adachi JD, Noseworthy MD, Maly MR. Efficacy of a biomechanically-based yoga exercise program in knee osteoarthritis: A randomized controlled trial. PLoS One. 2018 Apr 17;13(4):e0195653. doi: 10.1371/journal.pone.0195653. eCollection 2018. PMID 29664955

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M)
Started | 10 | 11 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants met the diagnostic criteria for clinical knee OA according to the American College of Rheumatology (Altman et al., 1986).
Groups:
- Total: Total of all reporting groups
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M) | Total
Number analyzed (Participants) | 10 | 11 | 10 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (5.6) | 63.7 (8.9) | 71.1 (9.3) | 66.7 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 10 | 31
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 11 | 10 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Lower Extremity Function
Description: The Lower Extremity Function Scale (LEFS) consists of 20 items, on an adjectival scale, that assess difficulty during mobility tasks ranging from transfers to running. The LEFS is scored from 0 to 80 with higher scores represent better self-reported physical function. It is reliable and valid in knee OA and has superior sensitivity to change compared to similar measures. The mean (95% confidence interval) difference score (follow-up score - baseline score) was computed for each of the three study arms.
Time Frame: Week 1 and Week 13
Measure: Mean (95% Confidence Interval); unit: Change in scores on a scale
Groups:
- Biomechanical Exercise (BE): The participants in this arm were asked to attend 3 group classes per week for 12 weeks at a local yoga studio taught by a certified yoga instructor. Four class times were offered per week. These classes included a warm-up, static poses shown to decrease knee joint loading, and a cool down including flexibility exercises. Measurements were obtained at baseline (before intervention) and at follow-up (following intervention).
- Traditional Exercise (TE): The participants in this arm were prescribed an aerobic and strengthening exercise program often prescribed to those with knee OA. The program included 15 minutes of walking per class, closed kinetic chain strengthening exercises on machines, and a cool down consisting of stretching. Participants were asked to come to class 3 times per week for 12 weeks. Certified Kinesiologists as well as student volunteers were available during all class times for program completion and progression. Measurements were obtained at baseline (before intervention) and at follow-up (following intervention).
- Meditation Control (M): The participants in this arm were asked to attend 3 meditation classes per week for 12 weeks taught by a certified yoga instructor with a specialization in meditation. These classes took place at an alternate area of the yoga studio to avoid contamination. Since it is known that exercise is beneficial for pain management and strengthening in knee OA, participants randomized to the control group were offered a free exercise pass following completion of the study. Measurements were obtained at baseline (before intervention) and at follow-up (following intervention).
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M)
Number analyzed (Participants) | 10 | 10 | 10
Change in scores on a scale | 10.6 [3.3 to 17.9] | 7.6 [-0.6 to 15.8] | -6.4 [-13.2 to 0.4]

2. Secondary Outcome: Change in Self-reported Knee Pain
Description: Change in self-reported knee pain was assessed with 3 valid and reliable questionnaires: the Knee injury and Osteoarthritis Outcome Score (KOOS), the Intermittent and Constant Osteoarthritis Pain (ICOAP) score, and the Numeric Pain Rating Scale (NPRS). The KOOS pain score represents a normalized score from 0 (extreme symptoms) to 100 (no symptoms). KOOS scores closer to 100 indicate fewer symptoms. The ICOAP consists of two sub-scales: constant pain (5 items) and intermittent pain (6 items). The score from each subscale represents a normalized score from 0 (no pain) to 100 (extreme pain). ICOAP scores closer to 0 indicate less pain. The NPRS pain score represents a score from 0 (no pain) to 10 (worst possible pain). NPRS ratings were provided following maximum isometric knee extensor exertions and flexor exertions. The mean (95% confidence interval) difference score (follow-up score - baseline score) was computed for each of the three study arms.
Time Frame: Week 1 and Week 13
Measure: Mean (95% Confidence Interval); unit: Change in scores on a scale
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M)
Number analyzed (Participants) | 10 | 10 | 10
Change in scores on a scale
  KOOS Pain | 21.5 [15.1 to 27.9] | 8.3 [-4.1 to 20.7] | -2.1 [-12.6 to 8.4]
  ICOAP Intermittent Pain | -23.7 [-30.9 to -16.5] | -14.3 [-23.4 to -5.2] | -4.2 [-16.7 to 8.3]
  ICOAP Constant Pain | -24.5 [-40.0 to -9.0] | -15.0 [-29.5 to -0.5] | -10.5 [-34.1 to 13.1]
  NPRS Extensor | -1.6 [-2.6 to -0.6] | -0.7 [-2.2 to 0.8] | 2.8 [0.1 to 5.5]
  NPRS Flexor | -0.9 [-2.3 to 0.5] | -0.3 [-1.9 to 1.3] | 2.3 [0.0 to 4.6]

3. Secondary Outcome: Change in Arthritis-related Self-efficacy
Description: The Arthritis Self-Efficacy Scale (ASES) measures arthritis-specific beliefs regarding perception of performance on certain tasks to cope with the disease. The ASES is measured using 20 questions on a 10-100 scale with respect to three main areas: pain management (5 questions), physical function (9 questions), and other symptoms (6 questions). Higher numbers indicate greater certainty that a participant can cope with a particular task as a consequence of their disease. The mean (95% confidence interval) difference score (follow-up score - baseline score) was computed for each of the three study arms.
Time Frame: Week 1 and Week 13
Measure: Mean (95% Confidence Interval); unit: Change in scores on a scale
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M)
Number analyzed (Participants) | 10 | 10 | 10
Change in scores on a scale | 0.2 [-4.4 to 4.8] | 2.6 [0.3 to 4.9] | 0.7 [-2.6 to 4.0]

4. Secondary Outcome: Change in Depression Status
Description: Depression was assessed with the Centre of Epidemiological Studies Depression (CES-D) Scale, a 20-item scale developed for the general population with emphasis on affect. Elements of affect include mood, guilt, worthlessness, helplessness, appetite, and sleep. The CES-D is scored from 0 to 60 with a score of 16 or higher indicating depression. The mean (95% confidence interval) difference score (follow-up score - baseline score) was computed for each of the three study arms.
Time Frame: Week 1 and Week 13
Measure: Mean (95% Confidence Interval); unit: Change in scores on a scale
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M)
Number analyzed (Participants) | 10 | 10 | 10
Change in scores on a scale | 1.0 [-4.6 to 2.6] | 1.0 [-3.5 to 1.5] | -3.6 [-9.5 to 6.2]

5. Secondary Outcome: Change in Frailty Status
Description: Frailty was assessed using the Edmonton Frail Scale (EFS). The EFS is a brief screening interview for older adults to assess frailty that is commonly used in both inpatient and outpatient settings. The scale covers 8 domains: cognition, general health status, functional independence, social support, medication use, nutrition, mood, continence, and functional performance (defined as performance on the Timed Up and Go [TUG] test). The test is scored out of 17, with higher scores indicating higher levels of frailty. The mean (95% confidence interval) difference score (follow-up score - baseline score) was computed for each of the three study arms.
Time Frame: Week 1 and Week 13
Measure: Mean (Full Range); unit: Change in scores on a scale
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M)
Number analyzed (Participants) | 10 | 10 | 10
Change in scores on a scale | 0.3 [-0.7 to 1.3] | -0.2 [-1.5 to 1.1] | -1.1 [-1.9 to -0.3]

6. Secondary Outcome: Change in Mobility Performance (Six-Minute Walk Test)
Description: Mobility performance was measured using the Six-Minute Walk Test. For this test, participants are instructed to walk as far as possible in 6 minutes. The distance covered in 6 minutes is recorded. This measure has produced reliable and valid data in persons with knee OA. The mean (95% confidence interval) difference in distance in metres (follow-up - baseline) was computed for each of the three study arms.
Time Frame: Week 1 and Week 13
Measure: Mean (95% Confidence Interval); unit: Change in metres
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M)
Number analyzed (Participants) | 10 | 10 | 10
Change in metres | 59.3 [22.5 to 96.0] | 54.0 [28.5 to 79.5] | 19.1 [-16.8 to 54.9]

7. Secondary Outcome: Change in Mobility Performance (40m Walk Test)
Description: Mobility performance was measured using the 40m Walk Test. This test measures the time taken to complete a fast-paced 40m walk. This measure has produced reliable and valid data in persons with knee OA. The mean (95% confidence interval) difference in time in seconds (follow-up - baseline) was computed for each of the three study arms.
Time Frame: Week 1 and Week 13
Measure: Mean (95% Confidence Interval); unit: Change in seconds
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M)
Number analyzed (Participants) | 10 | 10 | 10
Change in seconds | -3.9 [-7.4 to -0.3] | -2.9 [-5.0 to -0.8] | 4.0 [-9.9 to 17.9]

8. Secondary Outcome: Change in Mobility Performance (30-second Chair Stand Test)
Description: Mobility performance was measured using the 30-second Chair Stand Test. This test measures the number of times participants can rise and lower from a standard height chair, without using arm rests, in a 30-second period. This measure has produced reliable and valid data in persons with knee OA. The mean (95% confidence interval) difference in number (follow-up - baseline) was computed for each of the three study arms.
Time Frame: Week 1 and Week 13
Measure: Mean (95% Confidence Interval); unit: Change in number of sit-to-stand cycles
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M)
Number analyzed (Participants) | 10 | 10 | 10
Change in number of sit-to-stand cycles | 3.4 [2.0 to 4.8] | 2.5 [0.9 to 4.1] | 1.8 [0.3 to 3.3]

9. Secondary Outcome: Change in Mobility Performance (Timed Up and Go Test)
Description: Mobility performance was measured using the Timed Up and Go Test. This test measures the time taken to rise from a standard chair with arm rests, walk 3m, and return to a seated position. This measure has produced reliable and valid data in persons with knee OA. The mean (95% confidence interval) difference in time in seconds (follow-up - baseline) was computed for each of the three study arms.
Time Frame: Week 1 and Week 13
Measure: Mean (95% Confidence Interval); unit: Change in seconds
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M)
Number analyzed (Participants) | 10 | 10 | 10
Change in seconds | -1.3 [-2.3 to -0.3] | -0.3 [-1.0 to 0.4] | 0.2 [-1.2 to 1.6]

10. Secondary Outcome: Change in Mobility Performance (Stair Ascent)
Description: Mobility performance was measured using the Stair Ascent Test. For this test, the time taken to ascent nine stairs is recorded. The mean (95% confidence interval) difference in time in seconds (follow-up - baseline) was computed for each of the three study arms.
Time Frame: Week 1 and Week 13
Measure: Mean (95% Confidence Interval); unit: Change in seconds
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M)
Number analyzed (Participants) | 10 | 10 | 10
Change in seconds | -1.7 [-2.8 to -0.7] | -0.7 [-1.3 to -0.2] | 1.9 [-2.8 to 6.5]

11. Secondary Outcome: Change in Isometric Knee Extensor and Flexor Strength
Description: The peak torque developed during knee extension and flexion during a maximum voluntary isometric contraction was measured by use of a Biodex System 2 isokinetic dynamometer. The mean (95% confidence interval) difference in torque (follow-up - baseline) was computed for each of the three study arms. Data is presented as Nm/kg.
Time Frame: Week 1 and Week 13
Measure: Mean (95% Confidence Interval); unit: Change in Nm/kg
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M)
Number analyzed (Participants) | 10 | 10 | 10
Change in Nm/kg
  Knee Extensor Torque | 0.1 [0.0 to 0.2] | 0.0 [0.0 to 0.1] | 0.0 [-0.1 to 0.1]
  Knee Flexor Torque | 0.0 [-0.1 to 0.1] | 0.1 [0.0 to 0.2] | 0.0 [-0.1 to 0.1]

12. Secondary Outcome: Change in Isokinetic Knee Extensor and Flexor Power
Description: The peak isokinetic torque developed during knee extension and flexion at 25% resistance of their maximum voluntary isometric contraction was measured by use of a Biodex System 2 isokinetic dynamometer. The mean (95% confidence interval) difference in power (follow-up - baseline) was computed for each of the three study arms. Data is expressed in W/kg.
Time Frame: Week 1 and Week 13
Population: One participant in TE did not complete the power evaluation.
Measure: Mean (95% Confidence Interval); unit: Change in W/kg
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M)
Number analyzed (Participants) | 10 | 9 | 10
Change in W/kg | 0.3 [0.0 to 0.6] | 0.8 [0.3 to 1.3] | -0.1 [-0.4 to 0.2]

13. Secondary Outcome: Change in Grip Strength (Absolute)
Description: Peak grip strength was assessed using a Jamar hand dynamometer. The hand dynamometer was set to a fixed position and all values of grip force were expressed in kg. The mean (95% confidence interval) difference in absolute force (follow-up - baseline) was computed for each of the three study arms.
Time Frame: Week 1 and Week 13
Population: Note: only 9 participants were analyzed for the Left Side
Measure: Mean (95% Confidence Interval); unit: Change in kg
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M)
Number analyzed (Participants) | 10 | 10 | 10
Change in kg
  Right Side Grip Strength | 0.4 [-1.0 to 1.7] | -0.1 [-2.3 to 2.1] | 1.2 [-0.3 to 2.7]
  Left Side Grip Strength | 1.0 [-0.1 to 2.1] | -1.5 [-3.9 to 1.0] | 0.1 [-1.0 to 1.2]

14. Secondary Outcome: Change in Grip Strength (Relative)
Description: Peak grip strength was assessed using a Jamar hand dynamometer. The hand dynamometer was set to a fixed position and all values of grip force were expressed in kg/kg (grip force/body mass). The mean (95% confidence interval) difference in relative force (follow-up - baseline) was computed for each of the three study arms.
Time Frame: Week 1 and Week 13
Population: Note: only 9 participants were analyzed for the Left Side
Measure: Mean (95% Confidence Interval); unit: Change in kg/kg
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M)
Number analyzed (Participants) | 10 | 10 | 10
Change in kg/kg
  Right Side Normalized Grip Strength | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Left Side Normalized Grip Strength | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

15. Secondary Outcome: Change in Cardiovascular Fitness
Description: Cardiovascular fitness will be calculated using the YMCA submaximal cycle ergometry test. Predictions of VO2max will be made from heart rate (measured with a heart rate monitor) and load (Watts).
Time Frame: Intended to be collected on week 1 and week 13
Population: Data for this outcome measure were not collected.
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M)
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Change in Muscle and Fat Volume
Description: Muscle and fat volumes from magnetic resonance images will be segmented using a custom program. The images will be acquired using a • Iterative Decomposition of water and fat with Echo Asymmetry and Least-squares estimation (IDEAL) sequence on a 3.0T MR750 Discovery research-grade scanner.
Time Frame: Indented to be collected on week 1 and week 13
Population: Data for this outcome measure were not collected.
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M)
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Change in Cartilage Morphology
Description: Cartilage morphology will be assessed in open-sourced and custom programs. Sodium (23Na+) images and T2 mapping will be completed on the 3.0T MR750 DIscovery research-grade scanner. The mean (95% confidence interval) percent change from baseline to follow-up was computed for each of the three study arms.
Time Frame: Week 1 and Week 13
Measure: Mean (95% Confidence Interval); unit: % Change from Baseline to Follow-up
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M)
Number analyzed (Participants) | 7 | 6 | 9
% Change from Baseline to Follow-up
  T2 - Medial Femur | -3.7 [-13.5 to 6.0] | -1.0 [-9.2 to 7.1] | -1.3 [-9.4 to 6.8]
  T2 - Lateral Femur | 3.2 [-2.6 to 8.9] | -2.2 [-6.5 to 2.1] | -1.2 [-5.8 to 3.3]
  T2 - Medial Tibia | -1.8 [-11.8 to 8.3] | -3.0 [-8.5 to 2.5] | 3.9 [-5.0 to 12.7]
  T2 - Lateral Tibia | -1.9 [-10.9 to 7.1] | -0.7 [-13.6 to 12.2] | 7.5 [0.9 to 14.1]
  Volume - Medial Femur | -1.4 [-14.4 to 11.7] | -6.2 [-20.1 to 7.6] | -2.6 [-10.6 to 5.4]
  Volume - Lateral Femur | 2.4 [-2.2 to 6.9] | -5.0 [-13.2 to 3.2] | -0.4 [-7.2 to 6.5]
  Volume - Medial Tibia | 2.2 [-3.9 to 8.2] | 0.7 [-8.1 to 9.5] | -7.3 [-16.7 to 2.1]
  Volume - Lateral Tibia | 3.9 [-2.2 to 9.9] | 2.5 [-11.1 to 16.2] | 0.6 [-7.6 to 8.7]
  Thickness - Medial Femur | -2.6 [-10.9 to 5.7] | -1.9 [-9.0 to 5.1] | -3.1 [-11.7 to 5.5]
  Thickness - Lateral Femur | 0.2 [-2.4 to 2.8] | -3.4 [-10.2 to 3.3] | 2.1 [-3.0 to 7.2]
  Thickness - Medial Tibia | 2.0 [-1.0 to 5.0] | 0.7 [-3.6 to 4.9] | -5.4 [-9.7 to -1.0]
  Thickness - Lateral Tibia | 1.1 [-3.2 to 5.5] | 1.3 [-1.3 to 3.9] | -0.4 [-2.8 to 2.0]

18. Secondary Outcome: Change in Inflammatory Markers (IL6, TNF, IL10)
Description: Cytokines interleukin-6 (IL6), tumour necrosis factor (TNF), and interleukin-10 (IL10) are important markers of the inflammatory response. These markers will be assessed using standard blood draw and nasal swabs collected by a medical professional. The mean (95% confidence interval) difference in concentration in pg/ml (follow-up - baseline) was computed for each of the three study arms.
Time Frame: Week 1 and Week 13
Population: For IL10: n=6 (BE), n=8 (TE), n=6 (M)
Measure: Mean (95% Confidence Interval); unit: Change in pg/ml
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M)
Number analyzed (Participants) | 6 | 8 | 7
Change in pg/ml
  IL6 | -0.6 [-1.9 to 0.7] | 0.0 [-0.6 to 0.6] | 0.1 [-0.4 to 0.6]
  TNF | -3.4 [-9.4 to 2.7] | 0.3 [-0.8 to 1.3] | 0.3 [-1.9 to 2.5]
  IL10 | -11.9 [-44.4 to 20.6] | -2.6 [-5.0 to -0.1] | 1.2 [-0.5 to 2.9]

19. Secondary Outcome: Change in Inflammatory Markers (CRP)
Description: C-reactive protein (CRP) is an important marker of the inflammatory response. This markers will be assessed using standard blood draw and nasal swabs collected by a medical professional. The mean (95% confidence interval) difference in concentration in ug/ml (follow-up - baseline) was computed for each of the three study arms.
Time Frame: Week 1 and Week 13
Measure: Mean (95% Confidence Interval); unit: Change in ug/ml
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M)
Number analyzed (Participants) | 5 | 5 | 5
Change in ug/ml | 16.3 [-0.2 to 32.7] | -12.3 [-41.8 to 17.1] | -12.0 [-67.1 to 43.2]

ADVERSE EVENTS:
Arm/Group | Biomechanical Exercise (BE) | Traditional Exercise (TE) | Meditation Control (M)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/10

LIMITATIONS AND CAVEATS:
* The sample was statistically underpowered to detect all potential differences between and within groups
* This study involved only women thus limiting the generalizability

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No